CLINICAL TRIAL: NCT06029049
Title: Comparison of Intubation Conditions During Rapid Sequence Induction Obtained With Modified Time Principal Induction With a Standard Intubation Dose of Rocuronium Versus Succinylcholine : A Prospective Non-inferiority Randomized and Blind Trial
Brief Title: Comparison of Intubation Conditions During Rapid Sequence Induction Obtained With Modified Time Principal Induction With a Standard Intubation Dose of Rocuronium Versus Succinylcholine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Lauren Nakazawa, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-23-0468
Record Dates: First submitted 2023-08-22; First posted 2023-09-08 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified Time Principle Induction (MTPI) with rocuronium (Experimental)
  Interventions: Drug: Modified Time Principle Induction (MTPI) with rocuronium
- RSI with succinylcholine (Active Comparator)
  Interventions: Drug: RSI succinylcholine

INTERVENTIONS:
Drug: Modified Time Principle Induction (MTPI) with rocuronium — Participants will be induced using lidocaine 1 mg/kg IV, an opioid such a fentanyl (1-2 mcg/kg) IV, followed by 0.6 mg/kg IV rocuronium, and IV propofol with dosage at the discretion of the care team, administered within 10 seconds of rocuronium and the intubation will be performed with a C-MAC
  Arms: Modified Time Principle Induction (MTPI) with rocuronium
Drug: RSI succinylcholine — Participants will be induced as per routine care using lidocaine 1 mg/kg IV, an opioid such a fentanyl (1-2 mcg/kg) IV, propofol 1-2 mg/kg IV, and succinylcholine 1mg/kg IV, and the intubation will be performed with a C-MAC
  Arms: RSI with succinylcholine

SUMMARY:
The purpose of this study is to assess and compare conditions for tracheal intubation obtained with modified time principal induction with 0.6 mg/kg rocuronium and 1 mg/kg succinylcholine. Specifically, the investigators will be evaluating ease of laryngoscopy, vocal cord view, vocal cord opening, and movement of limbs and coughing during tracheal intubation in order to assess intubation conditions, to compare efficiency and success rate of tracheal intubation between two induction agents and to determine the rate of patient awareness during induction and post-operative recall of paralysis.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30kg/m2 or Mallampati class III or IV.
* Requiring general anesthesia and endotracheal intubation

Exclusion Criteria:

* Acute and chronic respiratory disorders, including Chronic obstructive pulmonary disease(COPD) and asthma.
* The American Society of Anesthesiologists (ASA) physical status classification > III.
* Patients requiring awake intubation.
* Pregnant women.
* Untreated ischemic heart disease.
* Patients requiring an induction dose of propofol < 1 mg/kg.
* Allergy to propofol, rocuronium, succinylcholine, or sugammadex.
* Patients with renal failure and unknown potassium (K+) level, or patients with K+ level > 5.0
* Personal history of malignant hyperthermia (MH), or family history of MH
* Patients with suspected or diagnosed neuromuscular disease, patients with burn injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Ease of laryngoscopy | During procedure (Between laryngoscope insertion to onset of ventilation (less than 7 minutes))
  Ease of laryngoscopy is scored categorically as easy (Jaw relaxed, no resistance to blade during laryngoscopy) , fair (Jaw not fully relaxed, some resistance to blade) or difficult (Poor jaw relaxation, active resistance by patient to laryngoscopy)
Position of vocal cords | During procedure (Between laryngoscope insertion to onset of ventilation (less than 7 minutes))
  Position of vocal cords is scored categorically as abducted, intermediate or closed
Movement of vocal cords | During procedure (Between laryngoscope insertion to onset of ventilation (less than 7 minutes))
  Movement of vocal cords is scored categorically as none , moving or closing
Number of participants who moved their limbs during intubation | During procedure (Between laryngoscope insertion to onset of ventilation (less than 7 minutes))
  none, slight or vigorous
number of participants who coughed during tracheal intubation | During procedure (Between laryngoscope insertion to onset of ventilation (less than 7 minutes))
  none, diaphragm or sustained (>10s)

SECONDARY OUTCOMES:
Number of participants for whom tracheal intubations were successful on the first attempt | 5 minutes after intubation and successful ventilation
Number of times tracheal intubations are attempted | 5 minutes after intubation and successful ventilation
Number of participants for whom tracheal intubations failed | After 3 failed intubation attempts (less than 7 minutes from start of intubation)
Airway view at the time of laryngoscopy as categorized by the modified Cormack-Lehane classification (before external manipulation) | from start of induction to 5 minutes of successful ventilation
  Data is reported categorically as follows 1(Full view of glottis),2a(Partial view of glottis), 2b(Only posterior extremity of glottis seen or only arytenoid cartilages), 3(Only epiglottis seen, none of glottis seen) and 4(Neither glottis nor epiglottis seen)
Satisfaction of providers with intubating conditions | from 5 minutes of successful ventilation
  Providers will answer yes or no for satisfaction
Heart Rate | from the start of induction drug administration to about 5 minutes after successful ventilation
Diastolic Blood Pressure | from the start of induction drug administration to about 5 minutes after successful ventilation
Systolic Blood Pressure | from the start of induction drug administration to about 5 minutes after successful ventilation
End-tidal carbon dioxide (CO2) | from the start of induction drug administration to about 5 minutes after successful ventilation
Oxygen saturation (SpO2) | from the start of induction drug administration to about 5 minutes after successful ventilation
Number of participants that had injury associated with intubation | within 24 hours after surgery
  Injury is defined as injury to dentition, lips, tongue, and pharyngeal bleeding.
Number of participants with muscle paralysis awareness prior to loss of consciousness as assessed by the Post Anesthesia Care Unit Survey of Modified Time Principle Induction | within 24 hours after surgery
Number of participants who had presence of sore throat as assessed by the score on the Post Anesthesia Care Unit Survey of Modified Time Principle Induction | within 24 hours after surgery
  This is scored from 0(no pain) to 10(worst pain)
Number of participants who had nausea as assessed by the score on the Post Anesthesia Care Unit Survey of Modified Time Principle Induction | within 24 hours after surgery
Number of participants who had vomiting as assessed by the score on the Post Anesthesia Care Unit Survey of Modified Time Principle Induction | within 24 hours after surgery
Overall patient satisfaction as assessed by the score on the Post Anesthesia Care Unit Survey of Modified Time Principle Induction | within 24 hours after surgery
  This is scored from 0(not satisfied) to 10(extremely satisfied)
Number of participants who had recollection of pain on induction | within 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Nakazawa, MD,MBA, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No